CLINICAL TRIAL: NCT02472743
Title: Light-based Therapy as a Novel Treatment for Digital Ulcers in Patients With Systemic Sclerosis
Brief Title: Light Treatment for Scleroderma Finger Ulcers
Acronym: DULight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Michael Hughes, Arthritis Research UK Clinical Research Fellow, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/196DERM
Record Dates: First submitted 2015-01-23; First posted 2015-06-16 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Scleroderma, Systemic; Ulcer
Keywords: Phototherapy
MeSH Terms: conditions — Scleroderma, Systemic; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Custom-built phototherapy lamp (Experimental): Custom-built phototherapy lamp:
  All participants will receive light treatment twice weekly for three weeks (or until ulcer/s healing) to one or both hands (both hands if ulcer/s present bilaterally).
  The participant will place their hand within the treatment area of the light-based device (total treatment area approximately 15cm2), aiming to centralise the digital ulcer/s to the centre of the treatment region.
  At each treatment study visit (visits 1-6 inclusive), the device will undergo a period of (automatic) calibration before use. All three wavelengths (red, infrared and blue) will be delivered simultaneously in combination, with the fluence of the device set at [3J/cm2] (treatment duration approximately 10 to 15 minutes).
  Interventions: Device: Custom-built phototherapy lamp

INTERVENTIONS:
Device: Custom-built phototherapy lamp — Described in the arm description
  Other Names: N/A: Custom built in house

SUMMARY:
Digital (finger) ulcers are common in patients with systemic sclerosis (SSc) and causes much pain and affects how patients use their hands. Our current treatments for digital ulcers are often not effective and have may have significant side effects (because they increase blood flow to the ulcer to try and help healing).

Light-based treatment has been successfully used to treat chronic diabetic, pressure and venous ulcers. The investigators wish to investigate whether light-based treatment is a safe and effective treatment for digital ulcers in patients with SSc.

DETAILED DESCRIPTION:
Study design This is an open pilot study: all participants will receive the light-based treatment (visits 1-6 inclusive). Ten participants with at least one digital ulcer (more than one digital ulcer may be assessed in the study if located on the same hand) will be recruited.

Justification of sample size There are no pilot data to inform a power calculation. Paired measurements on 10 participants gives 90% power to detect a clinically meaningful change in VAS of 2 points at the 5% significance level, provided that the observed standard deviation in paired differences is 1.7 or less. If the observed standard deviation is 2.0, this sample size gives 80% power to detect such a change at the stated significance level.

Methods of data collection

Study visits schedule Participants will attend a total of 8 study visits over two months. Light treatment will be administered twice weekly for three weeks (i.e. the first 6 study visits only). Follow-up visits will be at 1 month (visit 7) and 2 months (visit 8).

Preparation Participants will be asked to abstain from caffeine-containing drinks and from smoking for at least 4 hours prior to study. Sterile gauze and/or water may be used by the investigators (using gloves) to clean the surface of the wound of any debris that could potentially interfere with the light-based treatment.

Application of the light-based device to the digital ulcer Both the participant and investigators will wear appropriate safety goggles (as advised by Medical Physics at Salford Royal NHS Foundation Trust [SRFT]) at all times whilst the light-based device is in operation. The participant will place their hand within the treatment area of the light-based device (total treatment area approximately 15cm2), aiming to centralise the digital ulcer/s to the centre of the treatment region. The device will be controlled by a custom-built computer interface. At each study visit, the device will undergo a period of (automatic) calibration before use. All three wavelengths (red, infrared and blue) will be delivered simultaneously in combination, with the fluence of the device set at [3J/cm2] (treatment duration approximately 10 to 15 minutes). Performance data on the light-based treatment (including the total dose delivered and the performance of the LEDs will be recorded. In the event of catastrophic failure of the device (e.g. failure of multiple LEDs), the device will automatically shut down.

Participant and investigator assessment of feasibility Participant and the investigators opinion of the feasibility of light-based treatment will be recorded (at the end of the first and last treatment study visit).

Participant and investigator assessment of tolerability Participant and investigator opinion of the tolerability of light-based treatment will be recorded (at the end of the first and last treatment study visit).

Participant and investigator opinion Participant and investigator global assessments of the digital ulcer will be performed on a visual analogue scale (0-10, 10 being most severe) at each study visit. A clinical photograph (see immediately below) will be independently scored at a later date by another investigator.

Clinical Photography The Clinical Photography department at SRFT will take a photograph of the digital ulcer/s at the end of each study visit.

High-frequency ultrasound (HFUS) Will be performed immediately by the investigator after the light-treatment has been delivered and at the follow up visits. The investigator will perform two 'scans' along the short and long axis of the ulcer and use these to make measurements (basal and superficial width/length and volume).

Laser Doppler imaging (LDI) Will be performed by the investigator immediately before and directly after treatment (at the digital ulcer site and the corresponding contralateral arm position) at all visits to measure ulcer perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of SSc.
* Eighteen years of age or older at the time of recruitment.
* Able to give full informed consent.
* An active digital ulcer on any aspect of the finger/s (e.g. digital-tip or extensor)

Exclusion Criteria:

* Unable to give full informed consent.
* Serious infection of the digital ulcer e.g. osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety measured by the patient and operator opinion | Up to three weeks
Number of participants with adverse events as a measure of tolerability measured by the patient opinion | Up to three weeks

SECONDARY OUTCOMES:
Digital ulcer severity: participant and operator reported | Up to 8 weeks
  Up to 8 weeks
High-frequency ultrasound (HFUS) to measure digital ulcer dimensions | Up to 8 weeks
  Up to 8 weeks
Laser Doppler imaging (LDI) to measure perfusion to the digital ulcer | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hughes, MSc MRCP, Principal Investigator — The University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, Manchester, United Kingdom